CLINICAL TRIAL: NCT02521311
Title: A Randomized, Double-Blind, Parallel-Group, Placebo Controlled Trial to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of Clemastine Fumarate as a Remyelinating Agent in Acute Optic Neuritis
Brief Title: Assessment of Clemastine Fumarate as a Remyelinating Agent in Acute Optic Neuritis (ReCOVER)
Acronym: ReCOVER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-17428
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Optic Neuritis
Keywords: multiple sclerosis; eye pain; vision loss
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis; Eye Pain; Vision Disorders | interventions — Clemastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clemastine (Experimental): Participants will receive clemastine until 3 months and then will be off treatment until 9 month time point.
  Interventions: Drug: Clemastine
- Placebo (Placebo Comparator): Participants will receive placebo until 3 months and then will be off treatment until 9 month time point.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clemastine — 12mg (4mg 3x/day) clemastine for 7 days followed by 8mg clemastine (4mg 2x/day) until 3 months. Patients will be off treatment from 3-9 months and will be reevaluated at 9 months.
  Other Names: Tavist; Clemastine fumarate; Walhist
  Arms: Clemastine
Drug: Placebo — Equivalent placebo. 12mg (4mg 3x/day) placebo for 7 days followed by 8mg placebo (4mg 2x/day) until 3 months. Patients will be off treatment from 3-9 months and will be reevaluated at 9 months.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess clemastine as a remyelinating agent in patients with acute optic neuritis.The study will also evaluate the tolerability of clemastine, originally approved as first-generation antihistamine, in patients with optic neuritis. Study procedures will include assessments for evidence of remyelination in the anterior visual pathway and in the brain using electrophysiologic techniques and magnetic resonance imaging. If they are on one, patients in this study can remain on their standard disease modifying treatment during the course of the study. However, patients cannot participate in any other investigational new drug research study concurrently.

DETAILED DESCRIPTION:
Optic neuritis is an inflammatory, demyelinating disease of the optic nerve. It is most often characterized by visual loss or blurred vision along with dyschromatopsiaaccompanied by pain (especially with eye movement) and no demonstrable evidence of an alternate diagnosis such as ischemia or retinal disease. It can also be associated with a swollen optic disc (Optic Neuritis Study Group 1991, Hutchinson, W.M. 1976) and optic nerve enhancement on MRI (Kupersmith 2002).

Functional high-throughput screening for compounds that promote remyelination presents a major unmet need in the therapeutic arsenal for multiple sclerosis and other demyelinating conditions such as optic neuritis. Screening for myelin repair is problematic, as functional remyelination requires the presence of intact neuronal axons. Standard methods are not suited for high-throughput formats. We performed a detailed screen of over 1500 FDA approved small molecule drugs to identify agents that could be promising for remyelination. Engineered with conical dimensions, our micropillar technology permitted resolution of the extent and length of membrane wrapping from a single 2-dimensional image. Confocal imaging acquired from the base to the tip of the pillars allows for the fluorescence detection of concentric wrapping observed as "rings" of myelin membrane. The platform was formatted in 96-well plates, amenable to semi-automated random acquisition and automated detection and quantification. Upon initiating a screen of 1500 bioactive molecules, we identified Clemastine as a compound that potentially enhances oligodendrocyte differentiation and remyelination. We then validated this and other drugs in preclinical assays as well as in animal models of primary myelination and remyelination after inflammatory and chemical demyelination. Together, our findings illustrate the proof of concept for a novel high-throughput screening platform for potential regenerative therapeutics in MS (Chan JR et al. 2014).

This study is intended to assess for clinical evidence of remyelination using Clemastine Fumarate in patients with acute inflammatory injury causing demyelination of the anterior visual pathway as a consequence of acute demyelinating optic neuritis. The study is designed to assess tolerability and clinical efficacy of Clemastine using outcomes intended to assess for (a) adverse events and (b) recovery of myelin. This study is complementary to an earlier study evaluating clemastine in chronic demyelinated optic neuropathy and serves as part of a proof of concept program intended to evaluate methods for conducting remyelination trials in MS.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed or suspected to have an acute demyelinating optic neuritis in at least one eye within 3 weeks from the onset of any visual symptom other than pain
* Use of disease-modifying therapies is not a contraindication
* Use of appropriate contraception during the period of trial (women)
* Understand and sign the informed consent

Exclusion Criteria:

* Other major ophthalmologic diseases / concomitant ophthalmologic disorders (e.g. diabetes, macular degeneration, glaucoma, severe myopia, etc)
* Disc hemorrhages in the qualifying eye
* No light perception in qualifying eye
* Simultaneous bilateral optic neuritis
* Cotton wool spots in the qualifying eye
* Macular star in the qualifying eye
* History of significant cardiac conduction block
* History of cancer
* Suicidal ideation or behavior in 6 months prior to baseline
* Pregnancy, breastfeeding or planning to become pregnant
* Involved with other study protocols simultaneously without prior approval
* Concomitant use of any other putative remyelinating therapy as determined by the investigator
* Serum creatinine > 1.5 mg/dL; aspartate transaminase (AST), alanine transaminase (ALT), or alkaline phosphatase > 2 times the upper limit of normal
* History of drug or alcohol abuse within the past year
* Untreated B12 deficiency (as determined by B12 serological assessments and metabolites including methylmalonic acid (MMA) and homocysteine) or untreated hypothyroidism
* Clinically significant cardiac, metabolic, hematologic, hepatic, immunologic, urologic, endocrinologic, neurologic, pulmonary, psychiatric, dermatologic, allergic, renal, or other major diseases that, in the PI's judgment, may affect the interpretation of study results or patient safety
* History or presence of clinically significant medical illness or laboratory abnormality that, in the opinion of the investigator would preclude participation in the study.
* Positive for NMO antibody discovered within the first 2 weeks after randomization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in P100 latency on full-field visual evoked potential | baseline, 1 week, 1 month, 3 months, 9 months
  To evaluate the efficacy of clemastine relative to placebo for reducing P100 latencies on full field transient pattern reversal visual evoked potentials. Measure will be reported as difference in P100 latency from baseline to 9 months.
Change in low contrast visual acuity | baseline, 1 week, 1 month, 3 months, 9 months
  The second primary outcome is to measure the effectiveness of clemastine relative to placebo at improving patient performance on ETDRS low contrast visual acuity chart testing (2.5% black on white) during the recovery from an acute optic neuritis. Measure will be reported as difference in ETDRS score from baseline to 9 months.

SECONDARY OUTCOMES:
Change in retinal nerve fiber layer thickness on optical coherence tomography | baseline, 1 week, 1 month, 3 months, 9 months
  The primary outcome is to measure the effectiveness of clemastine relative to placebo at preventing the loss of retinal nerve fiber assessed via optical coherence tomography (OCT). Measure will be reported as difference in nerve fiber thickness between baseline and 9 months.
Radiological outcomes assessed by magnetic resonance imaging | baseline, 9 month
  To evaluate the efficacy of clemastine relative to placebo in increasing magnetization transfer ratios and myelin water fraction derived from magnetic resonance imaging of the brain during the period of exposure to active treatment. Measures will be reported as change between baseline and 9 months.
Expanded Disability Status Scale score | baseline, 9 months
  To evaluate the efficacy of Clemastine relative to placebo in reducing the EDSS score at 9 months.The EDSS is an ordinal scale used for assessing neurological impairment of MS based on a neurological examination. It consists of scores in each of seven functional systems (FS) and an ambulation score that are then combined to determine the EDSS [ranging from 0 (normal) to 10 (death due to MS)]. The FSs are the Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, and Cerebral functions. The FSs and EDSS steps will be assessed in a standardized manner. EDSS is a widely used and accepted instrument to evaluate disability status at a given time and longitudinally, to assess disability progression in clinical studies in MS.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Green, MD, MCR, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Mei F, Fancy SPJ, Shen YA, Niu J, Zhao C, Presley B, Miao E, Lee S, Mayoral SR, Redmond SA, Etxeberria A, Xiao L, Franklin RJM, Green A, Hauser SL, Chan JR. Micropillar arrays as a high-throughput screening platform for therapeutics in multiple sclerosis. Nat Med. 2014 Aug;20(8):954-960. doi: 10.1038/nm.3618. Epub 2014 Jul 6. PMID 24997607